CLINICAL TRIAL: NCT02401477
Title: Dual Therapy With High Doses of Ilaprazole and Amoxicillin for Helicobacter Pylori Infection; Studies From Korea
Brief Title: Dual Therapy With High Doses of Ilaprazole and Amoxicillin for Helicobacter Pylori Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DUMC-LYJ-ILA01
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Helicobacter Infections
Keywords: helicobacter pylori; ilaprazole; eradication; dual therapy; high dose therapy
MeSH Terms: conditions — Helicobacter Infections | interventions — ilaprazole; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ilaprazole + Amoxicillin (Experimental): Noltec(Ilaprazole) 10mg 4 tablets BID + Ildong-Amoxicillin 500mg 1capsule and 250mg 1capsule QID by oral for 14 days
  Interventions: Drug: Ilaprazole + Amoxicillin

INTERVENTIONS:
Drug: Ilaprazole + Amoxicillin — Ilaprazole 40mg BID, dosage form : delayed release tablet Amoxicillin 750mg QID, dosage form : capsule
  Other Names: Ilaprazole; Amoxicillin

SUMMARY:
This study assessed eradication rate of dual therapy with high doses of Ilaprazole 40mg BID and Amoxicillin 750mg QID for 14 days on Helicobacter pylori infection.

DETAILED DESCRIPTION:
The study performed to assess the eradication rate of H.pylori after 14 days treatment. The treatment is defined as those participants who confirmed on gastric or duodenal ulcer (including scar stage) or gastritis by endoscopy or the participants who received endoscopic treamtment for gastric polyp, gastric adenocarcinoma, confirmed to be H.pylori positive patients by the Biopsy or CLO test or Serological Diagnosis.

Patients administered Ilaprazole 40mg BID and Amoxicillin 750mg QID for 14days. The eradication rate on High dose dual therapy assessed by UBT test at Day 49±7.

ELIGIBILITY:
Inclusion Criteria:

* Subject who is confirmed on gastric or duodenal ulcer (including scar stage) by endoscopy or among the participants who received endoscopic treamtment for gastric polyp, gastric adenocarcinoma, confirmed to be H.pylori positive patients by the Biopsy, CLO test and Serological Diagnosis.
* Subject who fully understands conditions of clinical trial.
* Subject who agrees to participate and spontaneously sign the ICF

Exclusion Criteria:

* Known hypersensitivity to any component of Ilaprazole, Amoxicillin(Penicillin Antibiotics).
* Subjects who are taking contraindicated medications for experimental and concomitant drug.
* Administrated of PPI, antibiotic medication within 4 weeks prior to commencement of the study.
* Pregnant and/or lactating women
* Reproductive aged women not using contraception
* Uncontrolled diabetics
* Uncontrolled hypertension
* Uncontrolled liver dysfunction
* Uncontrolled kidney dysfunction
* Alcoholics
* Subjects with a history or possibility of digestive malignancy within 5 years
* Subjects with a history of gastrectomy or esophagectomy
* Subjects with hereditary diseases such as Galactose intolerance, Lapp lactose deficiency, glucose-galactose malabsorption.
* Infectious mononucleosis patients
* Subjects participating in a clinical trial before another trial wihin 30 days
* Inconsistence judged subject by researcher

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The eradication rate of H.pylori | Day 49±7
  The eradication rate of H.pylori after 14 days treatment is defined as those participants who confirmed on gastric or duodenal ulcer (including scar stage) or gastritis by endoscopy or the participants who received endoscopic treatment for gastric polyp, gastric adenocarcinoma, confirmed to be H.pylori positive patients by the Biopsy or CLO test or Serological Diagnosis.

SECONDARY OUTCOMES:
The number of patients with Adverse Events | Day 49±7

CONTACTS AND LOCATIONS:
Overall Officials: YoonJeong Lim, MD, PhD, Principal Investigator — DongGuk University
Locations (1):
- Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi-do, South Korea